CLINICAL TRIAL: NCT01103258
Title: FOAM-study Cost Minimization Study Comparing Surgery Versus Duplex Guided Foam Sclerotherapy of Varicose Veins: a Randomized Controlled Study
Brief Title: FOAM-study, Cost Minimization Study Comparing Surgery Versus Duplex Guided Foam Sclerotherapy of Varicose Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Dr A Sommer, Maastricht UMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 05-2-014; ZON MW 4636 (Other Grant/Funding Number: ZON MW)
Record Dates: First submitted 2010-04-06; First posted 2010-04-14 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Varicose Vein Disease
Keywords: Incompetence of the great saphenous vein.
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high ligation and stripping (Active Comparator): surgery consisting of high ligation in combination with long saphenous stripping
  Interventions: Procedure: high ligation and stripping (surgery)
- duplex guided foam sclerotherapy (Active Comparator): duplex guided foam sclerotherapy
  Interventions: Procedure: FOAM

INTERVENTIONS:
Procedure: high ligation and stripping (surgery) — surgery consisting of high ligation in combination with long saphenous stripping
  Arms: high ligation and stripping
Procedure: FOAM — duplex guided foam sclerotherapy
  Arms: duplex guided foam sclerotherapy

SUMMARY:
Varicose vein disease is a common health problem, which causes much discomfort to patients.

Nowadays treatment modalities for greater saphenous veins include surgery and duplex guided foam sclerotherapy. These are two equally accepted and applied treatments for the same patient population.

Choice of treatment often depends on the referral preference of the General Practitioner. Until now data are missing which treatment is more cost effective. The current proposal aims at comparing the effects, costs and patient preferences between duplex guided foam sclerotherapy and surgery in the treatment of greater varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* incompetence of great saphenous vein for minimal 20 cm
* life expectancy at least 3 years
* open and competent deep venous system
* willing to undergo both treatments

Exclusion Criteria:

* active ulcer
* signs of deep venous thrombosis with duplex
* incompetence of the deep venous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
cumulative probability of recurrent varicose vein within 24 months after treatment | 24 months

SECONDARY OUTCOMES:
quality of life (as measured by EuroQol-5D) | 24 months
patient preferences (as measured by conjoint analysis) | 24 months
direct Health care costs | 24 months
  materials, operation costs, personnel costs

CONTACTS AND LOCATIONS:
Overall Officials: A Sommer, MD PhD, Study Director — Maastricht UMC
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

REFERENCES:
- [Derived] Shadid N, Ceulen R, Nelemans P, Dirksen C, Veraart J, Schurink GW, van Neer P, vd Kley J, de Haan E, Sommer A. Randomized clinical trial of ultrasound-guided foam sclerotherapy versus surgery for the incompetent great saphenous vein. Br J Surg. 2012 Aug;99(8):1062-70. doi: 10.1002/bjs.8781. Epub 2012 May 25. PMID 22627969